CLINICAL TRIAL: NCT00884468
Title: Anxiety and Depression in Patients With Psoriatic Arthritis: Prevalence and Characteristics
Brief Title: Study Evaluating Anxiety and Depression in Patients With Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0881A5-4468
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Psoriatic Arthritis
Keywords: Anxiety and depression in patients with psoriatic arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with PsA that fulfill the eligibility criteria of the study

SUMMARY:
This is an epidemiological non-interventional study assessing the prevalence of anxiety and/or depression disorders in patients suffering from Psoriatic Arthritis (PsA) in Spain.

ELIGIBILITY:
Inclusion criteria:

* Patients both genders over 18 years old
* Patients with PsA diagnosis

Exclusion criteria:

* Patients with PsA that suffer from other rheumatologic diseases or non-concomitant rheumatologic diseases that the investigator considers not to be appropriate for the study.
* Patients with any medical or physical condition (cognitive damage or difficulties for understanding) that create difficulties for reading and completing the questionnaires described in the protocol.
* Patients that in the study period are taking part in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PsA from outpatient's surgery or primary health care centres
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of anxiety and/or depression disorders in patients suffering from PsA in Spain as measured by the Hospital Anxiety and Depression Scale (HAD) | 12 months

SECONDARY OUTCOMES:
To assess the relation between the PsA severity and the presence of anxiety and/or depression disorders in patients suffering from PsA in Spain. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Reus, Tarragona, Spain